CLINICAL TRIAL: NCT04511351
Title: Radiotherapy Combined With GDP (Gemcitabine, Cisplatin, Dexamethasone) Chemotherapy With or Without Chidamide in High-risk Early-stage Extranodal Nasal NK/T-cell Lymphoma
Brief Title: Radiotherapy Combined With GDP With or Without Chidamide in Stage I/II Extranodal Nasal NK/T-cell Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mei Dong, Director Physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMS lymphoma
Record Dates: First submitted 2020-08-10; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT+GDP+Chidamide (Experimental): IMRT followed by GDP chemotherapy with chidamide during radiation and chemotherapy phase
  Interventions: Drug: Chidamide
- RT+GDP (No Intervention): IMRT followed by GDP chemotherapy without chidamide during radiation and chemotherapy phase

INTERVENTIONS:
Drug: Chidamide — chidamide administration during radiation and chemotherapy phase in the study group
  Arms: RT+GDP+Chidamide

SUMMARY:
Currently, combined chemotherapy (CT) and radiation (RT) is recognized as the standard treatment for high-risk early-stage NKTCL. However, treatment failure occured in nearly 30% of patients receiving CRT and systemic failure are the most common failure form. Chidamide is a HADC inhibitor, which presents satisfactory efficacy in NKTCL especially in terms of improving durable remission time. In our previous study, IMRT followed by GDP was demonstrated effective in early-stage NKTCL. Therefore, we designed a prospective phase II clinical trial of IMRT followed by GDP with or without chidamide in patients with high-risk early-stage NKTCL.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of NKTCL with typical morphology and immunophenotype, according to the 2008 World Health Organization classification of lymphomas;
2. no prior radiotherapy or chemotherapy;
3. age ≥ 18 years;
4. ECOG performance status 0-2;
5. Ann Arbor stages I and II;
6. tumors primarily occurring in the upper aerodigestive tract;
7. at least one unfavorable prognostic factor (age > 60 years, B symptoms, elevated LDH, ECOG score 2, regional node involvement, and PTI);
8. at least one measurable lesion;
9. adequate hematological, hepatic, and renal functions; e.g., absolute neutrophil count ≥ 1.5 × 109/L, platelet count ≥ 80 × 109/L, total bilirubin ≤ 1.5 × upper limit of normal, alanine transaminase and aspartate transaminase ≤ 2 × upper limit of normal, and creatinine ≤ 1.5 mg/dl;
10. life expectancy of more than 3 months.

Exclusion Criteria:

1. Patients with advanced stage disease;
2. pregnancy or lactation;
3. any coexisting medical problems of sufficient severity to prevent full compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2014-08-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  Defined as the time from the date of study treatment until the earliest date of disease progression, as determined by radiographic disease assessment provided by an IRC, or death from any cause.

SECONDARY OUTCOMES:
Overall Survival | 2 years
  Defined as the time from the date of study treatment until death from any cause
Treatment response | 2 years
  Defined as the percentage of participants with a CR or PR as defined by revised response criteria for lymphoma (Cheson et al 2014)

CONTACTS AND LOCATIONS:
Overall Officials: Mei Dong, Principal Investigator — Cancer Hospital, Chinese Academy of Medical Scienses
Locations (1):
- National Cancer Center, Cancer Hospital, Chinese Academy of Medical Scienses, Beijing, Beijing Municipality, China